CLINICAL TRIAL: NCT04934566
Title: Comprehensive and Comparative Analysis of Venous Oxygen Saturation During ECMO Support: a Pilot Study
Brief Title: Venous Oxygen Saturation During ECMO Support
Acronym: ECMOxygen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019_58; 2020-A00505-34 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-03

CONDITIONS: Cardiogenic Shock
Keywords: Refractory cardiogenic shock; Extracorporeal life support; venous oxygen saturation; physiology
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Experimental): patients receiving temporary veno-arterial assistance whose weaning, or transfer to a heart transplant, or to long-term assistance or discontinuation is envisaged.
  Interventions: Other: ECMO flow

INTERVENTIONS:
Other: ECMO flow — Dynamic changes in ECMO flow and SvO2 measurement at the 3 different sites.

SUMMARY:
Extracorporeal veno-arterial membrane oxygenation" (ECMO-VA), are used to manage refractory cardiogenic shocks by replacing the failed "heart-lung" block. The Extracorporeal Life Support Organisation guidelines considers that the effectiveness of these techniques must be evaluated on the adequacy of tissue perfusion biomarker, of which is O2 saturation of venous blood found in the pulmonary artery using a Swan-Ganz catheter (SVO2) or in the superior vena cava/right atrium using a central venous catheter (ScVO2). During ECMO support, it can be also measured directly in the venous ECMO cannula (SmVO2).

However, due to the difference in tips locations of the venous cannula of ECMO-VA, the central venous catheter and the Swan-Ganz catheter, and rheological issues, the SmVO2, SVO2 and ScVO2 values obtained may be different.

Further we hypothesised that the level of admission flow may also affect the correlation between these different variables.

The aim of this experimental study is to investigate the concordance of the saturation of venous blood collected from these 3 measurement sites.

The primary objectives is to compare the concordance of ScVO2 and the SmVO2, the two more easily and systematically available variables

The secondary objectives were :

1. to evaluate the concordance of the 3 variables describing oxygen saturation
2. to analyse the primary objectives during prespecified and calibrated flow changes
3. analyse the association between these 3 variables with prognosis variables (Perfusion index, lactatemia, CO2 veno-arterial differences, SOFA score, SAPS II, successful weaning from the ECMO)
4. analyse in an ancilary study the concordance between SmVO2 measured using blood sample and the value obtained using a continuous monitoring of SVO2 through the circuit.

DETAILED DESCRIPTION:
Extracorporeal veno-arterial membrane oxygenation" (ECMO-VA), are used to manage refractory cardiogenic shocks by replacing the failed "heart-lung" block. The Extracorporeal Life Support Organisation guidelines considers that the effectiveness of these techniques must be evaluated on the adequacy of tissue perfusion biomarker, of which is O2 saturation of venous blood found in the pulmonary artery using a Swan-Ganz catheter (SVO2) or in the superior vena cava/right atrium using a central venous catheter (ScVO2). During ECMO support, it can be also measured directly in the venous ECMO cannula (SmVO2).

However, due to the difference in tips locations of the venous cannula of ECMO-VA, the central venous catheter and the Swan-Ganz catheter, and rheological issues, the SmVO2, SVO2 and ScVO2 values obtained may be different.

Further we hypothesised that the level of admission flow may also affect the correlation between these different variables.

The aim of this experimental study is to investigate the concordance of the saturation of venous blood collected from these 3 measurement sites.

The primary objectives is to compare the concordance of ScVO2 and the SmVO2, the two more easily and systematically available variables

The secondary objectives were :

1. to evaluate the concordance of the 3 variables describing oxygen saturation
2. to analyse the primary objectives during prespecified and calibrated flow changes
3. analyse the association between these 3 variables with prognosis variables (Perfusion index, lactatemia, CO2 veno-arterial differences, SOFA score, SAPS II, successful weaning from the ECMO)
4. analyse in an ancilary study the concordance between SmVO2 measured using blood sample and the value obtained using a continuous monitoring of SVO2 through the circuit.

ELIGIBILITY:
Inclusion Criteria:

* Weight >50 kg
* Veno-arterial ECMO with impending removal (for recovery, heart transplantation or LVAD/BIVAD implantation or support futility)
* Venous catheter tip positioned in the superior vena cava or right heart
* Arterial line for blood pressure monitoring
* Given informed consent

Exclusion Criteria:

* Pregnancy
* Absence of arterial line or central venous catheter
* Hemodynamic instability under ECMO support
* Malposition of ECMO venous canula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
the intraclass correlation coefficient (ICC) between SECMOO2, and ScVO2 in the initial assist condition of 2-3 L/min (after 30 minutes of stability) | after 30 minutes of stability in the initial assistance condition (condition 1)
  the intraclass correlation coefficient (ICC) between SECMOO2, and ScVO2 in the initial assist condition of 2-3 L/min (after 30 minutes of stability). Due to the importance of patient position, measurements will be standardized in supine position or with head of bed inclination less than 30% SVO2 measured on ECMO circuit and in patient's superior vena cava.

SECONDARY OUTCOMES:
ICC between SVO2 and SECMOO2 measured after 30 minutes of stability in the initial assist condition (2-3 L/min), in patients with a Swan-Ganz catheter | after 30 minutes of stability in the initial assistance condition (condition 1)
  The intraclass correlation between SVO2 and SECMOO2 measured after 30 minutes of stability in
ICC between ScVO2 and SVO2 measured after 30 minutes of stability | after 30 minutes of stability in the initial assistance condition (condition 1)
  Intracclass correlation between ScVO2 and SVO2 measured respectively in superior vena cava and pulmonary artery
Association between changes in SCVO2 and SECMOO2 measured at differents flow levels | More than 30 minutes of stability between each condition
  Changes in ScVO2 and SECMOO2 are measured at 4 differents conditions from Baseline (Condition 1). Those condictions will consist in 2 successive increaments in ECMO flow of 1000 ml each (Condition 2 and condition 3), followed by a return to the baseline ECMO Flow ( Condition 4)
Association between changes in SVO2 and SECMOO2 measured at differents flow levels | More than 30 minutes of stability between each condition
  Changes in ScVO2 and SECMOO2 are measured at 4 differents conditions from Baseline (Condition 1). Those condictions will consist in 2 successive increaments in ECMO flow of 1000 ml each (Condition 2 and condition 3), followed by a return to the baseline ECMO Flow ( Condition 4)
Association between each SVO2 derived variable with macrocirculatory, microcirculatory variables | More than 30 minutes of stability between each condition
  Association between ScVO2, SVO2, SECMOO2 with VIS score , Peripheral Perfusion Index and capillary refill time and arterial lactate

CONTACTS AND LOCATIONS:
Overall Officials: Mouhamed MOUSSA, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Service d'Anesthésie-Réanimation CCV Hôpital Cardiologique Centre Hospitalier et Universitaire de Lille, Lille, NORD, France